CLINICAL TRIAL: NCT01658397
Title: The Effect of Calorie Deprivation on Adipose Tissue Distribution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Pouneh K. Fazeli, MD, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2010P001066
Record Dates: First submitted 2012-08-01; First posted 2012-08-07 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Healthy
Keywords: Healthy subjects; Fasting; Weight loss
MeSH Terms: conditions — Fasting; Weight Loss | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fasting (Experimental): Ten day fast
  Interventions: Behavioral: Fasting

INTERVENTIONS:
Behavioral: Fasting — Ten day fast

SUMMARY:
In this study, we will be studying the effects of acute calorie deprivation (a 10-day fast) on bone marrow fat, other fat stores and bone parameters. We will be measuring changes in bone marrow fat using magnetic resonance spectroscopy and will use MRI to measure subcutaneous and visceral fat depots. Our hypothesis is that levels of bone marrow fat will increase after an acute fast.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 21-45 years
* 101-130% of ideal body weight as defined by the 1983 Metropolitan Life Insurance Height and Weight Tables
* Normal thyroid function
* Regular menses (women)
* Normal liver transaminases

Exclusion Criteria:

* Any disease known to affect bone metabolism, including untreated thyroid dysfunction, Cushing's syndrome, or renal failure
* Any medication known to affect bone metabolism -- including systemic steroids or immunosuppressants -- within three months of the study, excluding estrogen and progestins. Patients receiving depot medroxyprogesterone (Depo-Provera) will be excluded from participating for six months after their last injections. Bisphosphonates must have been discontinued for at least one year before participation
* Serum potassium <3.0 meq/L
* Pregnant and/or breastfeeding (women)
* Diabetes mellitus
* Active substance abuse, including alcohol
* Contraindications to MRI: cardiac pacemaker, metal implants, claustrophobia

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-09; Primary Completion 2014-07-21 (Actual); Study Completion 2014-07-21 (Actual)

PRIMARY OUTCOMES:
Change in Bone Marrow Adiposity over 10 day fasting period | Baseline, After 10 day fasting period
  Bone marrow adiposity will be measured before and after the 10 day fast using magnetic resonance spectroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Pouneh K Fazeli, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States